CLINICAL TRIAL: NCT02541812
Title: The Efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Obsessive Compulsive Disorder (OCD), a Pilot Study
Brief Title: The Use of Magnetic Brain Stimulation to Treat Obsessive Compulsive Disorder, a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2009:077
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2015-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Transcranial Magnetic Stimulation; Error processing
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): Ten sessions of 1Hz repetitive Transcranial Magnetic Stimulation of the dorsal anterior cingulate cortex in patients with obsessive compulsive disorder
  Interventions: Device: Transcranial Magnetic Stimulation
- Healthy Control Subjects (Active Comparator): One session of 1Hz repetitive Transcranial Magnetic Stimulation of the dorsal anterior cingulate cortex in healthy control individuals
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — A non-invasive method for brain stimulation

SUMMARY:
The purpose of this study is two-fold: first, to observe the effect of one session of repetitive transcranial magnetic stimulation (rTMS) on the error-prediction abilities of patients with obsessive compulsive disorder (OCD) as well as healthy individuals; and second, to observe the clinical effect of 10 sessions of rTMS in patients with OCD.

DETAILED DESCRIPTION:
A battery of cognitive tasks designed to selectively measure several aspects of anterior cingulate cortex (ACC) function, will be administered before and after one session of rTMS in all participants. The first neurocognitive session will be administered in a separate day from the rTMS session. The second neurocognitive session will be performed immediately after rTMS and in the same day. Participants will perform five tasks designed to test: error processing, error likelihood assessment, meta-memory, response inhibition, and affect recognition.

The rTMS paradigm will consist of four short trains of magnetic pulses which include 5 minutes of stimulation with 1Hz frequency (overall 1200 pulses in one session) with an intensity of 110% of each participant's motor threshold, and 2 minute intervals between the stimulation trains. Stimulation will be applied over the dorsal ACC (dACC) using a double-cone rTMS coil. dACC will be precisely targeted using neuronavigation software loaded a high resolution MRI of each subjects' brain.

OCD patients will go on to receive two weeks (10 sessions) of daily rTMS treatments using the same protocol described above.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed obsessive compulsive disorder
* Not currently receiving cognitive behavioural therapy
* Not currently on any medication or only taking one selective serotonin reuptake inhibitor (SSRI)

Exclusion Criteria:

* History of psychotic episodes
* History of neurological illness
* Previous head injury
* Active alcohol or substance abuse
* History of seizure disorders
* Currently pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Modirrousta, MD PhD FRCPC, Principal Investigator — University of Manitoba

REFERENCES:
- [Derived] Modirrousta M, Meek BP, Sareen J, Enns MW. Impaired trial-by-trial adjustment of cognitive control in obsessive compulsive disorder improves after deep repetitive transcranial magnetic stimulation. BMC Neurosci. 2015 Oct 9;16:63. doi: 10.1186/s12868-015-0205-z. PMID 26453446

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients | Healthy Control Subjects
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients | Healthy Control Subjects | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (12.1) | 29.5 (12.1) | 29.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 2 | 6 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Obsessive and Compulsive Symptom Severity (Yale-Brown Obsessive Compulsive Scale)
Description: Yale-Brown Obsessive Compulsive Scale. Minimum value = 0. Maximum value = 40. Higher scores indicate greater severity of obsessive and compulsive symptoms.
Time Frame: Recordings: baseline; after two weeks of rTMS
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Patients
Number analyzed (Participants) | 10
Percent change | -39.4 (15.4)

2. Secondary Outcome: Change in Post-error Slowing
Description: Post-error slowing (PES) is the difference in response time on trials following an error to trials following a correct response. Higher numbers indicate more post-error slowing (i.e. longer response times following an error trial compared to following a correct trial). The outcome measure is the change in PES from baseline to following one session of rTMS.
Time Frame: Recordings: baseline; after one session of rTMS
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Patients: One session of 1Hz repetitive Transcranial Magnetic Stimulation of the dorsal anterior cingulate cortex in patients with obsessive compulsive disorder
  Transcranial Magnetic Stimulation: A non-invasive method for brain stimulation
Arm/Group | Patients | Healthy Control Subjects
Number analyzed (Participants) | 10 | 10
ms | 1.4 (5.8) | -3.0 (4.8)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Patients | Healthy Control Subjects
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No